CLINICAL TRIAL: NCT02807246
Title: Effects of Probiotics on Neonatal Hyperbilirubinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Mehmet Mutlu, MD, Assoc. Prof., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014/115 24237859-120
Record Dates: First submitted 2016-06-08; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: Probiotic; Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Experimental: Breast milk+ Probiotics(Maflor®, Mamsel Pharmaceuticals, Turkey) The study group will be fed with probiotics at a dose of 1x109 CFU/day (Lactobacillus rhamnosus GG 109colony ). Probiotic is in a liquid drop form at a dose of 5 drops a day and is used orally for 10 days.
  Interventions: Biological: Maflor®, Mamsel Pharmaceuticals, Turkey
- Saline (Active Comparator): Active Comparator: Breast milk+five drops of saline The control group will be given Breast milk without the addition of probiotics
  Interventions: Other: drops of saline

INTERVENTIONS:
Biological: Maflor®, Mamsel Pharmaceuticals, Turkey — Dietary Supplement: Probiotics probiotics at a dose of 1x109 CFU/day. (Maflor®, Lactobacillus rhamnosus GG 109 CFU, Mamsel Pharmaceuticals, Turkey)
  Other Name: Maflor®
  Arms: Probiotic
Other: drops of saline — Dietary Supplement: Breast milk +drops of saline
  Arms: Saline

SUMMARY:
This study was designed as a prospective controlled study to investigate the effects of probiotic support started immediately after birth on newborn jaundice in breastfed babies born by normal spontaneous vaginal delivery.

DETAILED DESCRIPTION:
Objectives: Enterohepatic circulation of bilirubin imposes an extra burden of approximately 30% on total serum bilirubin levels. Intestinal microflora is the main factor affecting enterohepatic circulation. This study investigated the effects of probiotic support started immediately after birth on neonatal hyperbilirubinemia in babies born by normal spontaneous vaginal delivery and breastfed only.

Methods: A total of 150 healthy term newborns were included in the study and allocated in the study and control groups. Immediately after birth, newborns in the study group received probiotic in liquid drop form (Maflor® drops containing Lactobacillus Rhamnosus GG 109 Colony Forming Units(CFU), Mamsel Pharmaceuticals, Turkey), at a dose of 5 drops a day orally for 10 days. Newborns in the control group received 5 drops of saline solution per day orally, instead. In addition to routine biochemical examinations;serum bilirubin levels in the cord blood, and blood samples of the newborns on the 3rd, 5th and 10th days of birth were measured in all subjects in both groups. Defecation frequency was recorded for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* A total of 150 full-term (gestational age ≥37 - <42 weeks) normal spontaneous vaginal delivery healthy newborns
* Birth weight between the 10th-90th percentiles
* Fed by breast milk only

Exclusion Criteria:

* Newborns with familial hematologic disorders
* Having signs of hemolysis due to blood group incompatibilities
* Bleeding into closed spaces due to birth trauma complications (e.g. cephalohematoma)
* Suspected or documented neonatal infection such as chorioamnionitis, intrauterine infection, sepsis and urinary tract infection
* Perinatal and neonatal hypoxia
* Having thyroid dysfunction, respiratory distress or insufficiency, metabolic and thermoregulatory dysfunction, hemodynamic instability and congenital heart disease
* Maternal phenobarbital usage history during the last month of the pregnancy
* Having venous hematocrit (Htc) levels≥65%

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Effect of Probiotic Support on Serum Bilirubin Levels | Change from birth to ten days of life
  The effect of probiotic support on serum bilirubin levels during the first 10 days were measured and results were given as mg/dL.

SECONDARY OUTCOMES:
Defecation frequency | Change from birth to ten days of life
  Number of defecation frequency releated to treatment was evaluated and counted as times/a day.

CONTACTS AND LOCATIONS:
Overall Officials: Yakup Aslan, Study Chair — Division of Neonatology, Karadeniz Technical University Faculty of Medicine, Trabzon, Turkey

IPD SHARING:
Plan to Share IPD: Undecided